CLINICAL TRIAL: NCT01181596
Title: NICU-TECH RM9L-RS Probe ME Feasibility Study
Status: Terminated | Type: Observational
Why Stopped: Images not adequate to visualize catheter penetration or obtain measurements
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: NICU-TECH RM9L-RS
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-06

CONDITIONS: Neonates
Keywords: neonates and infants, from the 23-week gestational (0.5 kg); up to a 6 month old born at term (7 kg), for whom the PIV,; PAC, UAC, UVC or PICC catheter insertion is medically; indicated.
MeSH Terms: conditions — Atrial Premature Complexes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: observational ultrasound: Collection of image data with the ultrasound probe.

SUMMARY:
Use of a new ultrasound device designed for babies to look at the catheters in veins and arteries as well as the blood vessel itself. An observational study to assess the the clinicians perception of the ultrasound image quality as a tool to detect catheters in vessels.

DETAILED DESCRIPTION:
The intent of the study is to confirm the maximum penetration of the NICU-Tech RM9L-RS probe. The investigators collected images on patients with PIV (Peripheral Intra Venous)/PAC (Peripheral Arterial Catheter) and central line catheters. The investigators collected images of deep vessel structures for offline processing to improve NICU-Tech algorithms for vessel segmentation.

ELIGIBILITY:
Inclusion Criteria:

* Neonates that are 23 gestational weeks at birth (and greater than 500 grams) to a 6 month old born infant at term (maximum weight 7 kg) who already have one or more lines placed (PIV/PAC/UVC/UACs/PICC) as part of their medical care. NO INFANT WILL HAVE A LINE PLACE FOR THE PURPOSE OF THIS STUDY

Exclusion Criteria:

* Neonates that are less than 23 gestational weeks at birth
* Neonates that are 23 gestational weeks at birth but are less than 500 grams in weight
* Patients weighing more than 7 kg.-Patients older than 6 months

Ages: 23 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates and infants, from the 23-week gestational (0.5 kg) up to a 6 month old born at term (7 kg), for whom the PIV, PAC, UAC, UVC or PICC catheter insertion is medically indicated.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Kim, MD, Principal Investigator — UCSD Medical Center
Locations (1):
- UCSD Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational study where recruitment took place in the Neonatal Intensive Care Unit. Enrollment period of June 2010 - November 2011.
Pre-assignment Details: If participants health worsens prior to assignment they were excluded from the study.
Groups:
- Ultrasound Probing: Ultrasound probing to guide catheter placement
Period: Overall Study
Arm/Group | Ultrasound Probing
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects that underwent an ultrasound scan during the study
Arm/Group | Ultrasound Probing
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.5 (.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Participants That Fulfilled All Study Procedures.
Description: Acquisition of basic images and video were obtained from study participants who already have one or more catheters in place.
Time Frame: 1 day (day of procedure)
Population: Study participants who have one or more catheters in place.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Observational Ultrasound
Number analyzed (Participants) | 31
Participants | 31

2. Primary Outcome: Vessel Penetration of NICU-Tech RM9L-RS Probe
Description: The algorithmic depth of vessel penetration will be collected.
Time Frame: 1 day (day of procedure)
Population: Images were not adequate to visualize catheter penetration, or to obtain measurements.
Arm/Group | Ultrasound Probing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1.5 years
Arm/Group | Ultrasound Probing
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

LIMITATIONS AND CAVEATS:
Enrollment was stopped early/terminated, study development stopped and no results were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days